CLINICAL TRIAL: NCT03134612
Title: Comparison Between Ondansetron 8 mg and Lidocain 40 mg in Preventing Pain Due to Propofol Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aries Perdana, Consultant, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes005
Record Dates: First submitted 2017-04-24; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: General Anesthesia With Propofol
Keywords: lidocain; ondansetron; pain; propofol
MeSH Terms: conditions — Pain | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Ondansetron (Active Comparator): Ondansetron 8mg (2mg/cc) was given intravenously via a 20 G vein canula
  Interventions: Drug: Ondansetron 8 mg
- Lidocain (Active Comparator): Lidocain 40mg (20mg/cc + 2cc of normal saline) was given intravenously via a 20 G vein canula
  Interventions: Drug: Lidocain 40 mg

INTERVENTIONS:
Drug: Ondansetron 8 mg
  Arms: Ondansetron
Drug: Lidocain 40 mg
  Arms: Lidocain

SUMMARY:
This study aims to compare the effectivity between ondansetron 8 mg and lidocain 40 mg in preventing pain due to propofol injection

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study. Non-invasive blood pressure (NIBP) monitor, ECG and pulse-oximeter was set on the subjects in the operation room. After a tourniquet made from NIBP cuff were inflated, subjects were given either Ondansetron 8 mg or Lidocain 20 mg intravenously, then the tourniquet was set off. Hemodynamic data was recorded. Propofol 1 mg/kg of body weight (BW) injection was given. Verbal rating scale was used to measure pain at 0 s, 5 s and 30 s. Data was analyzed using Statistical Package for the Social Sciences (SPSS), for numeric data using uni-variate analysis and bi-variate analysis. Significant value is p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-65 years old
* Subjects were planned to undergo general anesthesia with propofol
* Subjects with Body Mass Index (BMI) 18-35 kg/m2
* Subjects with American Society of Anesthesiologists (ASA) physical status of I-II
* Subjects with signed informed consent.

Exclusion Criteria:

* Subjects with allergies to propofol, lidocain, ondansetron
* Subjects with massive cardiac disorder
* Subjects with cardiac rhythm disorder with or without treatment
* Subjects with unstable hemodynamic
* Subjects with contraindication to propofol, lidocain, ondansetron
* Subjects with intubation and ventilation difficulty
* Subjects with decreased consciousness, seizure history or head injury
* Subjects with analgesic treatment history
* Subjects with pregnancy.

Drop out criteria:

* Subjects with allergic reactions induced by propofol, lidocain, ondansetron
* Uncooperative subjects
* Subjects in emergency
* Subjects with difficult vein access in the dorsum manus
* Subjects with infection and/or inflammation in the planned intravenous cannulation location.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The Degree of pain due to Propofol Injection | Day 1
  The degree of pain due to propofol injection was measured at 0 second, 15 seconds, 30 second, using verbal rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Aries Perdana, Consultant, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marik PE. Propofol: therapeutic indications and side-effects. Curr Pharm Des. 2004;10(29):3639-49. doi: 10.2174/1381612043382846. PMID 15579060
- [Background] Jalota L, Kalira V, George E, Shi YY, Hornuss C, Radke O, Pace NL, Apfel CC; Perioperative Clinical Research Core. Prevention of pain on injection of propofol: systematic review and meta-analysis. BMJ. 2011 Mar 15;342:d1110. doi: 10.1136/bmj.d1110. PMID 21406529
- [Background] Tan CH, Onsiong MK. Pain on injection of propofol. Anaesthesia. 1998 May;53(5):468-76. doi: 10.1046/j.1365-2044.1998.00405.x. PMID 9659020
- [Background] Johnson RA, Harper NJ, Chadwick S, Vohra A. Pain on injection of propofol. Methods of alleviation. Anaesthesia. 1990 Jun;45(6):439-42. doi: 10.1111/j.1365-2044.1990.tb14328.x. PMID 2200299
- [Background] Macario A, Weinger M, Truong P, Lee M. Which clinical anesthesia outcomes are both common and important to avoid? The perspective of a panel of expert anesthesiologists. Anesth Analg. 1999 May;88(5):1085-91. doi: 10.1097/00000539-199905000-00023. PMID 10320175
- [Background] Ye JH, Mui WC, Ren J, Hunt TE, Wu WH, Zbuzek VK. Ondansetron exhibits the properties of a local anesthetic. Anesth Analg. 1997 Nov;85(5):1116-21. doi: 10.1097/00000539-199711000-00029. PMID 9356111
- [Background] Lee SK. Pain on injection with propofol. Korean J Anesthesiol. 2010 Nov;59(5):297-8. doi: 10.4097/kjae.2010.59.5.297. Epub 2010 Nov 25. No abstract available. PMID 21179288
- [Background] Massad IM, Abu-Ali HM, Abu-Halaweh SA, Badran IZ. Venous occlusion with lidocaine for preventing propofol induced pain. A prospective double-blind randomized study. Saudi Med J. 2006 Jul;27(7):997-1000. PMID 16830018
- [Background] Picard P, Tramer MR. Prevention of pain on injection with propofol: a quantitative systematic review. Anesth Analg. 2000 Apr;90(4):963-9. doi: 10.1097/00000539-200004000-00035. PMID 10735808
- [Background] Mangar D, Holak EJ. Tourniquet at 50 mm Hg followed by intravenous lidocaine diminishes hand pain associated with propofol injection. Anesth Analg. 1992 Feb;74(2):250-2. doi: 10.1213/00000539-199202000-00014. PMID 1731546
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] Tramer MR, Reynolds DJ, Moore RA, McQuay HJ. Efficacy, dose-response, and safety of ondansetron in prevention of postoperative nausea and vomiting: a quantitative systematic review of randomized placebo-controlled trials. Anesthesiology. 1997 Dec;87(6):1277-89. doi: 10.1097/00000542-199712000-00004. PMID 9416710
- [Background] Paventi S, Santevecchi A, Ranieri R. Efficacy of a single-dose ondansetron for preventing post-operative nausea and vomiting after laparoscopic cholecystectomy with sevoflurane and remifentanil infusion anaesthesia. Eur Rev Med Pharmacol Sci. 2001 Mar-Apr;5(2):59-63. PMID 11863320
- [Background] Azimaraghi O, Aghajani Y, Molaghadimi M, Khosravi M, Eslami K, Ghadimi F, Movafegh A. Ondansetrona reduz a dor da injecao de etomidato: estudo randomico controlado. Braz J Anesthesiol. 2014 May-Jun;64(3):169-72. doi: 10.1016/j.bjan.2013.06.014. Epub 2014 Mar 7. No abstract available. Portuguese. PMID 25456475
- [Background] Ambesh SP, Dubey PK, Sinha PK. Ondansetron pretreatment to alleviate pain on propofol injection: a randomized, controlled, double-blinded study. Anesth Analg. 1999 Jul;89(1):197-9. doi: 10.1097/00000539-199907000-00035. PMID 10389803
- [Background] Zahedi H, Maleki A, Rostami G. Ondansetron pretreatment reduces pain on injection of propofol. Acta Med Iran. 2012;50(4):239-43. PMID 22592573
- [Background] Powell RM, Buggy DJ. Ondansetron given before induction of anesthesia reduces shivering after general anesthesia. Anesth Analg. 2000 Jun;90(6):1423-7. doi: 10.1097/00000539-200006000-00032. PMID 10825334
- [Background] Yeh HM, Chen LK, Lin CJ, Chan WH, Chen YP, Lin CS, Sun WZ, Wang MJ, Tsai SK. Prophylactic intravenous ondansetron reduces the incidence of intrathecal morphine-induced pruritus in patients undergoing cesarean delivery. Anesth Analg. 2000 Jul;91(1):172-5. doi: 10.1097/00000539-200007000-00032. PMID 10866907
- [Background] Kyriakides K, Hussain SK, Hobbs GJ. Management of opioid-induced pruritus: a role for 5-HT3 antagonists? Br J Anaesth. 1999 Mar;82(3):439-41. doi: 10.1093/bja/82.3.439. PMID 10434832
- [Background] Ye JH, Ponnudurai R, Schaefer R. Ondansetron: a selective 5-HT(3) receptor antagonist and its applications in CNS-related disorders. CNS Drug Rev. 2001 Summer;7(2):199-213. doi: 10.1111/j.1527-3458.2001.tb00195.x. PMID 11474424
- [Background] Golparvar M, Saghaei M, Saadati MA, Farsaei S. Effect of ondansetron on prevention of post-induction hypotension in elderly patients undergoing general anesthesia: A randomized, double-blind placebo-controlled clinical trial. Saudi J Anaesth. 2015 Oct-Dec;9(4):365-9. doi: 10.4103/1658-354X.159455. PMID 26543450
- [Background] Reddy MS, Chen FG, Ng HP. Effect of ondansetron pretreatment on pain after rocuronium and propofol injection: a randomised, double-blind controlled comparison with lidocaine. Anaesthesia. 2001 Sep;56(9):902-5. doi: 10.1046/j.1365-2044.2001.02059-6.x. PMID 11531681
- [Background] Bolton CM, Myles PS, Carlin JB, Nolan T. Randomized, double-blind study comparing the efficacy of moderate-dose metoclopramide and ondansetron for the prophylactic control of postoperative vomiting in children after tonsillectomy. Br J Anaesth. 2007 Nov;99(5):699-703. doi: 10.1093/bja/aem236. Epub 2007 Aug 21. PMID 17715139
- [Background] Deegan R. Ondansetron: pharmacology of a specific 5HT3-receptor antagonist. Am J Med Sci. 1992 Dec;304(6):373-8. doi: 10.1097/00000441-199212000-00009. No abstract available. PMID 1456277
- [Background] Brill S, Middleton W, Brill G, Fisher A. Bier's block; 100 years old and still going strong! Acta Anaesthesiol Scand. 2004 Jan;48(1):117-22. doi: 10.1111/j.1399-6576.2004.00280.x. PMID 14674982
- [Background] van Zundert A, Helmstadter A, Goerig M, Mortier E. Centennial of intravenous regional anesthesia. Bier's Block (1908-2008). Reg Anesth Pain Med. 2008 Sep-Oct;33(5):483-9. doi: 10.1016/j.rapm.2008.04.011. PMID 18774520
- [Background] Rosenberg PH, Heavner JE. Multiple and complementary mechanisms produce analgesia during intravenous regional anesthesia. Anesthesiology. 1985 Jun;62(6):840-2. No abstract available. PMID 4003822
- [Background] Shevchenko Y, Jocson JC, McRae VA, Stayer SA, Schwartz RE, Rehman M, Choudhry DK. The use of lidocaine for preventing the withdrawal associated with the injection of rocuronium in children and adolescents. Anesth Analg. 1999 Apr;88(4):746-8. doi: 10.1097/00000539-199904000-00011. PMID 10195516
- [Background] Memis D, Turan A, Karamanlioglu B, Kaya G, Pamukcu Z. The prevention of propofol injection pain by tramadol or ondansetron. Eur J Anaesthesiol. 2002 Jan;19(1):47-51. doi: 10.1017/s0265021502000078. PMID 11913803
- [Background] Mahler SA, Massey G, Meskill L, Wang H, Arnold TC. Can we make the basilic vein larger? maneuvers to facilitate ultrasound guided peripheral intravenous access: a prospective cross-sectional study. Int J Emerg Med. 2011 Aug 25;4:53. doi: 10.1186/1865-1380-4-53. PMID 21867495
- [Background] Groothuis JT, van Vliet L, Kooijman M, Hopman MT. Venous cuff pressures from 30 mmHg to diastolic pressure are recommended to measure arterial inflow by plethysmography. J Appl Physiol (1985). 2003 Jul;95(1):342-7. doi: 10.1152/japplphysiol.00022.2003. Epub 2003 Apr 4. PMID 12679358
- [Background] Flaherty SA. Pain measurement tools for clinical practice and research. AANA J. 1996 Apr;64(2):133-40. PMID 9095685
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] McCrirrick A, Hunter S. Pain on injection of propofol: the effect of injectate temperature. Anaesthesia. 1990 Jun;45(6):443-4. doi: 10.1111/j.1365-2044.1990.tb14329.x. PMID 2200300
- [Background] Aubrun F, Paqueron X, Langeron O, Coriat P, Riou B. What pain scales do nurses use in the postanaesthesia care unit? Eur J Anaesthesiol. 2003 Sep;20(9):745-9. doi: 10.1017/s0265021503001212. PMID 12974598
- Available data/document: Textbook — https://sydney.edu.au/medicine/pmri/pdf/Acute-pain-management-scientific-evidence-third-edition.pdf — Assessment and measurement of pain and its treatment. In: Macintyre PE SD, Schug SA, Visser EJ, Walker SM, editors. Acute pain management: scientific evidence. Melbourne: Australian and New Zealand College of Anaesthetists and Faculty of Pain Medicine; 2010.p. 35-43
- Available data/document: Textbook — http://accessanesthesiology.mhmedical.com/book.aspx?bookID=413 — Candido KD, Winnie AP. Intravenous regional block for upper & lower extremity surgery. In: Hadzic A, editor. Textbook of regional anesthesia and acute pain management. New York: McGraw-Hill; 2007. p. 565-78